CLINICAL TRIAL: NCT02675023
Title: A Randomized, Open-label, Two-arm, Parallel Group, Single Dose Study to Assess the Pharmacokinetics and Safety of M923 Administered Via Auto-injector or Prefilled Syringe, in Healthy Subjects
Brief Title: Assessment of Pharmacokinetics and Safety of M923 Administered Via Auto-injector or Prefilled Syringe, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Momenta Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 911501
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2017-04

CONDITIONS: Healthy
MeSH Terms: interventions — Adalimumab

ARMS (2):
- Auto-injector (AI) (Experimental): M923 administered via AI
  Interventions: Biological: M923
- Prefilled syringe (PFS) (Experimental): M923 administered via PFS
  Interventions: Biological: M923

INTERVENTIONS:
Biological: M923 — Recombinant human immunoglobulin G subclass 1 (IgG1) monoclonal antibody specific for human tumor necrosis factor-alpha (TNF-α)
  Other Names: Adalimumab

SUMMARY:
This study will assess the pharmacokinetic (PK) and safety of a single 0.8 mL (40 mg) subcutaneous (SC) dose of M923 administered via an auto-injector (AI) or a prefilled syringe (PFS) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 55 years, inclusive
2. Healthy participants as determined by pre-study medical history, physical examination, vital signs and 12-lead electrocardiogram (ECG)
3. Participants with clinical laboratory test results that are not clinically significant and are acceptable to the investigator at screening and admission to the study site (Day -1)
4. Participants with a body weight between 60.0 kg and 100.0 kg and a body mass index between 18.5 kg/m2 and 34.9 kg/m2, inclusive
5. Healthy male participants must be willing to comply with the contraception restrictions for this study.

   -Male participants with non-pregnant female partners of childbearing potential should avoid conception of a child during the study (up to Day 71 post-dose) and for 90 days thereafter.
6. Healthy female participants must have a negative pregnancy test at screening and on admission to the study site (Day -1), must not be lactating and must be using an acceptable method of contraception throughout the study and for 30 days after study completion, or be of non-childbearing potential.

   -Non-pregnant female partners of male participants who are of childbearing potential should use an effective form of contraception.
7. Participants who have smoked ≤10 cigarettes or 3 cigars or 3 pipes/day for at least 3 months prior to screening and are willing to comply with smoking restrictions during residency at the study site
8. Participants who are able to understand and provide written informed consent including signature on an informed consent form (ICF) approved by an Ethics Committee (EC)/ Institutional Review Board (IRB)
9. Participants who have provided written authorization for use and disclosure of protected health information
10. Participants who agree to abide by the study schedule and dietary restrictions and to return for the required assessments

Exclusion Criteria:

1. History and/or current presence of clinically significant angioedema, or eczematous dermatitis that requires prescription medication, clinically significant hypersensitivity, or severe allergic reactions (either spontaneous or following IP administration), also including known or suspected clinically relevant drug hypersensitivity to any components of the IP or comparable drugs, including latex
2. Active or latent tuberculosis or who have a history of TB.
3. History of invasive and/or active systemic fungal infections or other severe opportunistic infections, including recurrent or clinically significant chronic local fungal infections
4. A serious infection within 6 months prior to investigational product (IP) administration and/or an infection within 2 weeks of screening or during the screening period unless resolved completely within 2 weeks of admission to the study site on Day -1
5. Herpes zoster infection in the last year or more than 2 herpes zoster infections in his/her lifetime
6. Frequent chronic or recurrent infections (defined as >3 a year requiring prescribed treatment)
7. Previous use of adalimumab, HUMIRA®, or another recombinant human monoclonal antibody
8. Intake of any investigational drug in another study within 30 days (or 5 half-lives, whichever is greater) prior to intake of IP in this study or have received the last dose of a study drug more than 30 days ago (or 5 half-lives, whichever is greater) but who are on extended follow-up, or planned intake of an investigational drug (other than for this study) during the course of this study
9. History of alcohol abuse in the year preceding the screening visit, or history of excess alcohol consumption.
10. Known history of opioid or cocaine drug abuse or any other drug abuse in the past year or positive tests for drugs of abuse or alcohol at screening or admission to the study site (Day -1)
11. Donation of blood or blood products (eg, plasma, platelets) within 30 days prior to IP administration
12. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), dietary supplements or herbal medication during the 2 weeks prior to IP administration or longer if the medication has a long half-life. Use of any medication deemed necessary by the participant's physician to treat or prevent any medical condition, paracetamol/acetaminophen ≤3 g/day and use of vitamins at daily recommended doses is allowed; for female volunteers, oral birth control and hormone replacement therapy is allowed
13. History of or existing congestive heart failure
14. History of or existing signs or symptoms of demyelinating disease such as optic neuritis and/or multiple sclerosis
15. History of any cancer including lymphoma, leukemia, skin cancer or cervical carcinoma in situ
16. Impaired liver function
17. History of immunodeficiency (including those participants with a positive test for human immunodeficiency virus [HIV] I and II at screening) or other clinically significant immunological disorders, or auto-immune disorders, (eg, rheumatoid arthritis, lupus erythematosus, scleroderma, psoriasis)
18. Positive test for anti-citrullinated protein antibodies at screening
19. Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological (including pancytopenia, aplastic anemia, or blood dyscrasia), metabolic (including known diabetes mellitus), lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders as judged by the investigator
20. Received a live vaccine within 12 weeks prior to admission to the study site (Day -1) or plan to receive a live vaccine during the study (up to and including Day 71)
21. Volunteers who are vegans or have medical dietary restrictions
22. Volunteers who cannot communicate reliably with the investigator
23. Volunteer is a family member or employee of the investigator or study site staff or study team

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 603 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve from 0 to infinity | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
  Area under the concentration-time curve in serum from time zero (predose) extrapolated to infinity [AUC(0-inf)]
Pharmacokinetics: Area under the concentration-time curve from 0 to 336 hours | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, and 15
  Area under the concentration-time curve in serum from time zero (predose) to 336 hours postdose [AUC(0-336)]
Pharmacokinetics: Maximum concentration in serum (Cmax) | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71

SECONDARY OUTCOMES:
Pharmacokinetics: Serum M923 concentration up to Day 71 | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Area under the concentration-time curve in serum from time zero (predose) to 1200 hours postdose [AUC(0-1200)] | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, and 50
Pharmacokinetics: Area under the concentration-time curve in serum from time zero (predose) to time of the last quantifiable concentration [AUC(0-last)] | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Time of maximum concentration in serum [tmax] | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
  Obtained directly from the observed concentration versus time data
Pharmacokinetics: Terminal rate constant (λ z) | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Terminal half-life (t½) | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Apparent volume of distribution (Vz/F) | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Apparent systemic clearance after extravascular dosing (CL/F) | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Area under the concentration-time curve extrapolated from time "t" to infinity [% AUCex] | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Pharmacokinetics: Area under the serum concentration-time curves from time zero (predose) to time "t" [AUC(0-t)] by which >20.0% of participants have developed neutralizing antidrug antibody [nADA] | Within 90 minutes pre-dose; and post-dose at 8 hours, and Day 2, 3, 4, 5, 6, 7, 9, 11, 15, 22, 29, 40, 50, and 71
Non-serious and serious adverse events (SAEs) | Throughout the study period of approximately 8 months
Incidence of injection site reactions | Throughout the study period of approximately 8 months
Clinically significant changes in Vital signs | Throughout the study period of approximately 8 months
Number of participants with new clinically significant findings from the physical examination | Throughout the study period of approximately 8 months
  Physical examination will be done on the following body systems: general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological.
Clinically significant changes in Twelve-lead electrocardiogram (ECG) | Throughout the study period of approximately 8 months
Clinically significant changes in laboratory results | Throughout the study period of approximately 8 months
Clinically significant changes in clinical chemistry | Throughout the study period of approximately 8 months
Clinically significant changes in urinalysis | Throughout the study period of approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: John Caminis, MD, Study Director — Shire
Locations (2):
- QOPK Phase 1 Clinic, Overland Park, Kansas, United States
- QLON Phase 1 Clinic, London, United Kingdom